CLINICAL TRIAL: NCT04498637
Title: Attitudes Towards Disability of Nursing and Physiotherapy Students
Status: Completed | Type: Observational
Sponsor: University of Extremadura (Other)
Collaborators: University of Cadiz (Other)
Responsible Party: Principal Investigator, Elisa María Garrido Ardila, PHD, University of Extremadura
Other Study IDs: POR-2017
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Disability Physical; Disabilities Multiple; Disability Hearing; Disability, Vision; Disability, Intellectual
Keywords: Physiotherapy students; Nursing students; Disability; Attitude
MeSH Terms: conditions — Vision Disorders; Intellectual Disability; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physiotherapy students: Students enrolled in the Physiotherapy Bachelor´s Degree of the University of Cadiz, Spain
  Interventions: Other: 'Attitudes towards people with disability Scale'
- Nursing students: Students enrolled in the Nursing Bachelor´s Degree of the University of Cadiz, Spain
  Interventions: Other: 'Attitudes towards people with disability Scale'

INTERVENTIONS:
Other: 'Attitudes towards people with disability Scale' — The scale 'Attitudes towards people with disability' was completed by the participants. This scale allows the analysis of the attitudes towards disability trough a score whose lower values indicate a more negative attitude and higher values indicate more positive attitudes.

SUMMARY:
The general objective of this study is to know the attitude towards people with disability of Nursing and Physiotherapy students in the University of Cadiz. This is a descriptive, correlational, transversal and synchronous study.

DETAILED DESCRIPTION:
Attitudes determine our behaviour to some extent. Health professionals should have a global perspective of disability. They must provide treatment to people with disability and care for them, but also should accept them with no judgements or discrimination. The general objective of this study is to know the attitude towards people with disability of Nursing and Physiotherapy students in the University of Cadiz. Method: This is a descriptive, correlational, transversal and synchronous study. A total of 200 students participate in the study (91 from the Bachelor's Degree in Nursing and 109 from the Bachelor's Degree in Physiotherapy). The 'Attitudes towards people with disability Scale' was used.

ELIGIBILITY:
Inclusion Criteria:

* Students from the Physiotherapy Bachelor´s Degree of the university of Cadiz
* Students from the Nursing Bachelor´s Degree of the university of Cadiz, Campus of Jerez de la Frontera and Cadiz

Exclusion Criteria:

* None

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students enrolled in the Physiotherapy or Nursing Bachelor´s Degree of the University of Cadiz during the academic year of 2017/2018
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Attitude towards disability | Through study completion, an average of 11 months
  The 'Attitudes towards people with disabilities scale' (G form) is the assessment tool used (Verdugo M., Jenaro C. y Arias B., 1994) to assess the attitude that students from Physiotherapy and Nursing in the University of Cadiz have. This scale allows the analysis of the attitudes towards disability trough a score whose lower values indicate a more negative attitude and higher values indicate more positive attitudes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cadiz, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No